CLINICAL TRIAL: NCT03841370
Title: Tooth Crown Discoloration Caused by Endodontic Treatment: Cross-sectional Clinical Study
Brief Title: Tooth Crown Discoloration Caused by Endodontic Treatment
Status: Completed | Type: Observational
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, Professor, Federal University of Pelotas
Other Study IDs: FUPel
Record Dates: First submitted 2018-11-19; First posted 2019-02-15 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Endodontically Treated Teeth; Root Canal Infection; Tooth Discoloration
MeSH Terms: conditions — Tooth, Nonvital; Tooth Discoloration | interventions — Endodontics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- endodontic: The color of anterior (incisors and canines) and posterior (premolar) teeth treated at a private clinic in the city of Pelotas will be evaluated. Data will be collected regardless of technique, treatment time and sealer used.
  The ΔE00 will be evaluated using the measurements obtained in the homologous tooth (without endodontic treatment) versus the measurement obtained from the tooth treated endodontically.
  The values of ΔE00 obtained for each sealer, cut and time will be analyzed by multifactorial analysis to verify associations of the outcomes with the ΔE00.
  Interventions: Procedure: endodontic treatment

INTERVENTIONS:
Procedure: endodontic treatment — Color measurements of endodontically treated teeth (incisors, canines or premolar) will be collected regardless of technique, treatment time and sealer used.

SUMMARY:
The color change of endodontically treated teeth is a common concern in clinical practice. The objective of this study will be to evaluate, in vivo, the color change (ΔE00) caused by endodontic treatment. A observational retrospective study will be conducted to evaluate the ΔE00 of anterior (incisors and canines) and posterior (premolar) teeth treated at a private clinic, regardless of technique, treatment time and sealer used. In this study the ΔE00 will be evaluated using the measurements obtained in the homologous tooth (without endodontic treatment) versus the measurement obtained from the tooth treated endodontically. The values of ΔE00 obtained for each sealer, cut and time will be analyzed by multifactorial analysis to verify associations of the outcomes with the ΔE00.

DETAILED DESCRIPTION:
This cross-sectional clinical study will evaluate the color difference (∆E00), and CIELAB coordinates (L*, a*, and b*) of endodontic treated teeth in the 3 conditions (baseline, homologous tooth versus ≤ 1 month after tooth endodontic treatment); (baseline, homologous tooth versus > 1 to 12 months after tooth endodontic treatment); (baseline, homologous tooth versus > 12 up to 5 years after tooth endodontic treatment). The following pairs of variables will be considered in the comparisons: filling material (AH Plus and Endofill/Fillcanal/MTA Fillapex); cut at cervical level (dental cervix and 2mm in the apical direction); and location tooth (anterior and posterior teeth).

The response variables will include the color difference (∆E00), estimated by the CIEDE2000 color difference metric (ΔE00) obtained from readings made on the homologous tooth of the endodontic treated (baseline) and tooth endodontic treated (after) with a spectrophotometer.

All individuals who came to a private dental clinic between January 2010 and December 2018 and who received endodontic treatment will be considered for participation in this study. The following inclusion criteria will be used to evaluate and enroll potential participants: individuals at least 18 years old; who received anterior or posterior (pre-molar) endodontic treatment and who present homologous tooth with pulp vitality and at least 1/3 of the remaining coronary, without endodontic treatment, intraradicular retentor or crown making dental color assessment impossible. Besides, will be excluded questionnaires filled incorrectly or lack of data regarding, the day, month and year of endodontic treatment finish, sealer used, the pulp condition at the time of the first consultation (irreversible pulpitis or pulpal necrosis) and periapical radiography, obtained with the use of radiographic positioner, preserved and with a clear image. All individuals who agree to participate in the study will sign a consent form based on the Declaration of Helsinki, after receiving information about the study objectives, risks, and benefits associated with the alternative treatment options and procedures. One examiner will be trained and calibrated prior to data collection. Kappa statistics will be used to assess intra-examiner reliability. Clinical, radiographic and color information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* endodontically treated tooth, without intraradicular retainer and fixation;
* presence of homologous tooth to that treated, with pulp vitality and at least 1/3 of the crown;
* correctly patient's file showing the endodontic treatment day, the endodontic filler used, the pulp condition at the first consultation, and periapical radiography, obtained with the use of a radiographic positioner, preserved and with a clear apical image

Exclusion Criteria:

* dental elements submitted to retreatment;
* files with insufficient data, and absence of quality periapical radiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent endodontic treatment and who presented the homologous tooth without endodontic treatment in order to perform a color comparison measurement.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Color alteration | ranging from 1 month to 5 years after endodontic treatment.
  Color alteration (CIEDE2000 color difference metric - ΔE00) will be evaluated using the measurements obtained in the homologous tooth (without endodontic treatment) versus the measurement obtained from the tooth treated endodontically.

CONTACTS AND LOCATIONS:
Overall Officials: Noéli Boscato, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil